CLINICAL TRIAL: NCT04179786
Title: An Open-label, Single Arm, Single Center Clinical Study In Healthy Subjects to Qualify an In-house Reference Standard Batch of Sci-B-Vac™
Brief Title: A Study to Qualify an In-house Reference Standard Batch of Sci-B-Vac™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SciB018
Record Dates: First submitted 2019-10-07; First posted 2019-11-27 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B
Keywords: SciB018; Prophylactic vaccine; Sci-B-Vac™; HepB vaccines; Phase 4; pre-S1; pre-S2; Surface antigen
MeSH Terms: conditions — Hepatitis B | interventions — Pre-S vaccine

STUDY DESIGN:
Intervention Model Description: This study was an open-label, single arm study. No control groups were deemed necessary since this was a phase IV trial for which the goal, set according to the European Pharmacopeia 1056, was to achieve 95% SPR after the third vaccination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sci-B-Vac™ (Other): Single arm study in healthy volunteers who had never been vaccinated with any hepatitis B vaccine and who were seronegative for antibodies to HBsAg, HBc and HBs at baseline.
  Interventions: Biological: Sci-B-Vac™

INTERVENTIONS:
Biological: Sci-B-Vac™ — Sci-B-Vac™ is a recombinant Hepatitis B vaccine, produced by SciVac Israel Ltd under good manufacturing practices (GMP). It contains the 3 surface antigens of the Hepatitis B virus: HBs, pre-S1 and pre-S2. Each 1 ml dose contains sterile 10 μg Hepatitis B virus surface antigens. It is formulated for intramuscular injection supplied in single use vials containing 1ml suspension.

SUMMARY:
Each Sci-B-Vac™ lot to be released to the market is tested in comparison to a reference batch,which has to be tested in a human clinical trial. This study was conducted by SciVac Ltd. to to evaluate the immunogenicity and explore the immune kinetics of Sci-B-Vac™ in support of its qualification as new reference standard which according to the European Pharmacopeia (Ph.Eur. 1056) should elicit ≥ 95% seroprotection rate (SPR) of Hepatitis B surface (HBs) antibody concentrations ≥ 10 milli-International Units (mIU) per ml in young, healthy adult subjects.

DETAILED DESCRIPTION:
This study was a post-marketing, open-label, single arm study in healthy volunteers who had never been vaccinated with any hepatitis B vaccine and were seronegative to HBsAg, Hepatitis B core (HBc) and HBs antibodies. This study consisted of three periods: screening period (up to 1 month prior to first vaccination), treatment (Day 1 to month 6), and post-vaccination follow-up period (months 6 -12). Immunogenicity endpoints were examined one month after the first injection and at every month until month 6, then at months 7, 9 and 12. The primary safety endpoint was the frequency, severity, and duration of adverse events, including clinically-significant laboratory abnormalities after administration of Sci-B-Vac™.

Statistical Methods: A total of 92 subjects were recruited into the study. Subjects who fully complied with the study protocol, had no inclusion/exclusion criteria violation and who early terminated the study but reached the primary endpoint prior to withdrawal (modified intention-to-treat (mITT) population) were included in the final population for statistical analysis. mITT population was defined as the subset of the ITT set, which consisted of all enrolled subjects who were vaccinated at least once with Sci-B-Vac™ and had at least one post-vaccination follow-up visit, fully complied with the protocol and had no violation of the inclusion/exclusion criteria. Eligible subjects were followed for a total duration of 12 months.

Significance Level: The overall significance level for this study was 5% using two-tailed tests. Sample size determination was performed under the following assumptions:

The primary endpoint for the study was the SPR, defined as the proportion of subjects with HBs antibody titer ≥10 mIU/ml by month 7 (i.e. one month after the third immunization with Sci-B-Vac™). Subjects terminated early from the study for any reason at any time and who met the primary endpoint were included.

In compliance with the European Pharmacopeia, the SPR threshold was set at ≥ 95%. Based on a 9% margin of non-inferiority, the study was considered successful if the lower bound of the 95.0% exact confidence interval (CI) was 86.0% or more (lower non-inferiority limit) by month 7.

The secondary objective of the study was to explore kinetics of immune response induced by Sci-B-Vac™ based on serial immunogenicity measurements.

Demographic and baseline data as well as disease prognostic factors, medical history and prior medications were summarized for the mITT population,For continuous variables, descriptive statistics (number [n], mean, standard deviation (SD), standard error, median, minimum, and maximum) were provided. For categorical variables, subject counts and percentages were provided.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females 20 - 40 years of age.
2. Subjects who provided written informed consent to participate in the study.
3. Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
4. No clinically-significant abnormalities in hematology, blood chemistry, or urinalysis lab tests at Screening.
5. Women of child-bearing potential had to practice an acceptable method of birth control or practice abstinence during the study period or be surgically sterilized, from Screening visit throughout the vaccination phase and for 28 days after the last injection and agree to undergo repeated pregnancy tests.
6. Subjects had to be able to understand the requirements of the study and willing to comply with the requirements of the study.

Exclusion Criteria:

1. Known history of significant medical disorder, which in the investigator's judgment contraindicates administration of the vaccine or may interfere with the subject's compliance or the interpretation of study assessment parameters.
2. Any clinically-significant abnormality upon physical examination or in the clinical laboratory tests at Screening visit.
3. Treatment with immune suppressive agents.
4. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
5. History of Hepatitis B virus (HBV) infection or confirmed exposure to HBV
6. Previous vaccination against Hepatitis B.
7. Positive for HBsAg, anti-HBs antibodies, anti-HBc antibodies, anti-HCV (hepatitis C virus) antibodies or anti- HIV antibodies.
8. Drug abuse
9. Known hypersensitivity or allergy to any component of the study vaccine.
10. Body mass index (BMI) < 18.5 or ≥ 30 kg/m2.
11. Known concomitant disease or any other medical condition that is considered by the investigator likely to interfere with the subject's compliance or the interpretation of study assessments.
12. Any acute illness (e.g. acute infection) within 48 hours prior to the first study drug administration that is considered of significance by the Principal Investigator.
13. Female subjects: pregnant, lactating or planning a pregnancy.
14. Any confirmed or suspected immunosuppressive or immunodeficient condition.
15. Receipt of blood or immunoglobulin transfusion six months prior to the first vaccine dose and during the course of the trial.
16. Unwilling or unable (in the judgment of the investigator) to comply with all the requirements of the protocol.
17. Participate in another clinical trial within 3 months prior to first vaccination (calculated from the previous study's last dosing date).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, MD, Study Director — TASMC Clinical Research Center (CRC)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atsmon J, Machluf N, Yayon-Gur V, Sabbah C, Spaans JN, Yassin-Rajkumar B, Anderson DE, Popovic V, Diaz-Mitoma F. Rapid and high seroprotection rates achieved with a tri-antigenic Hepatitis B vaccine in healthy young adults: Results from a Phase IV study. Vaccine. 2021 Feb 22;39(8):1328-1332. doi: 10.1016/j.vaccine.2020.12.050. Epub 2021 Jan 13. PMID 33451780

RESULTS

PARTICIPANT FLOW:
Groups:
- Sci-B-Vac™: Single arm study in healthy volunteers who had never been vaccinated with any hepatitis B vaccine and who were seronegative for antibodies to HBsAg, HBc and HBs at baseline.
  Sci-B-Vac™ is a recombinant Hepatitis B vaccine, produced by SciVac Israel Ltd under good manufacturing practices. It contains the 3 surface antigens of the Hepatitis B virus: HBs, pre-S1 and pre-S2. Each 1 ml dose contains sterile 10 μg Hepatitis B virus surface antigens. It is formulated for intramuscular injection supplied in single use vials containing 1ml suspension.
Period: Overall Study
Arm/Group | Sci-B-Vac™
Started | 91
Completed | 83
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Arm/Group | Sci-B-Vac™
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.24 (4.79)
Age, Customized [Count of Participants; unit: Participants]
  Between 20 and 30 years | 75
  Between 31 and 40 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 91
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Israel | 91

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Rate Achieved One Month After the Third Immunization With Sci-B-Vac™.
Description: SPR (% of subjects ≥ 10 mIU/mL) one month after immunization with Sci-B-Vac™ at months 0, 1 and 6 was calculated by measuring the HBs antibody titers using Cobas™ e601 anti-HBs assay. Subjects who received at least one Sci-B-Vac™ dose and early terminated from the study for any reason at any time while having HBs antibody concentrations ≥ 10 mIU/ml were considered among those who met the endpoint.
Time Frame: Month 7 (i.e. one month after the third immunization with Sci-B-Vac™)
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac™
Number analyzed (Participants) | 83
Participants | 83

2. Secondary Outcome: Seroprotection Rates Achieved Monthly During Treatment and Then at Month 7, 9 and 12 During Follow-up
Description: The endpoint for the study was the SPR, defined as the percentage of subjects with HBs antibody titer ≥10 mIU/ml. The Cobas™ e601 anti-HBs assay was used to assess the HBs antibody titer.
Time Frame: At one month after the first injection, and then at every month until month 7 inclusive and at months 9 and 12.
Population: The immunogenicity results presented here were obtained through analyses performed on the modified intent-to-treat (ITT) analysis set. This set consisted of all enrolled subjects who were vaccinated at least once with Sci-B-Vac™ at least one post vaccination follow-up visit, fully comply with the study protocol, had no violation of any of the inclusion/exclusion criteria and did not demonstrate an anamnestic response after the 1st administration of Sci-B-Vac™.
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac™
Number analyzed (Participants) | 88
Participants
  Month 1 | 50
  Month 2: number analyzed (Participants) | 86
  Month 2 | 79
  Month 3: number analyzed (Participants) | 86
  Month 3 | 85
  Month 4: number analyzed (Participants) | 84
  Month 4 | 83
  Month 5: number analyzed (Participants) | 83
  Month 5 | 82
  Month 6: number analyzed (Participants) | 83
  Month 6 | 82
  Month 7: number analyzed (Participants) | 83
  Month 7 | 83
  Month 9: number analyzed (Participants) | 83
  Month 9 | 83
  Month 12: number analyzed (Participants) | 84
  Month 12 | 84

3. Secondary Outcome: Percentage of Subjects With HBs Antibody Titer ≥100 mIU/ml at Each Timepoint
Description: The outcome was the proportion of subjects with HBs antibody titer ≥100 mIU/ml. The Cobas™ e601 anti-HBs assay was used to assess the HBs antibody titer.
Time Frame: At one month after the first injection, and then at every month until month 7 inclusive and at months 9 and 12.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Sci-B-Vac™
Number analyzed (Participants) | 88
Participants
  Month 1 | 32
  Month 2: number analyzed (Participants) | 86
  Month 2 | 66
  Month 3: number analyzed (Participants) | 86
  Month 3 | 70
  Month 4: number analyzed (Participants) | 86
  Month 4 | 71
  Month 5: number analyzed (Participants) | 83
  Month 5 | 70
  Month 6: number analyzed (Participants) | 83
  Month 6 | 70
  Month 7: number analyzed (Participants) | 83
  Month 7 | 81
  Month 9: number analyzed (Participants) | 83
  Month 9 | 80
  Month 12: number analyzed (Participants) | 84
  Month 12 | 77

4. Secondary Outcome: Geometric Mean Concentration (GMC) as Determined by HBs Antibody Titers
Description: The Cobas™ e601 anti-HBs assay was used to assess the HBs antibody titer.
Time Frame: At one month after the first injection, and then at every month until month 7 inclusive and at months 9 and 12.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/ml
Arm/Group | Sci-B-Vac™
Number analyzed (Participants) | 88
mIU/ml
  Month 1 | 1.49 [0.36 to 6.12]
  Month 2: number analyzed (Participants) | 86
  Month 2 | 358.62 [201.03 to 639.75]
  Month 3: number analyzed (Participants) | 86
  Month 3 | 413.59 [249.11 to 686.68]
  Month 4: number analyzed (Participants) | 84
  Month 4 | 379.06 [234.43 to 612.93]
  Month 5: number analyzed (Participants) | 83
  Month 5 | 343.89 [213.79 to 553.16]
  Month 6: number analyzed (Participants) | 83
  Month 6 | 300.30 [187.94 to 479.85]
  Month 7: number analyzed (Participants) | 83
  Month 7 | 6799.87 [4216.64 to 10965.66]
  Month 9: number analyzed (Participants) | 83
  Month 9 | 4170.86 [2610.57 to 6663.71]
  Month 12: number analyzed (Participants) | 84
  Month 12 | 2281.08 [1426.95 to 3646.49]

ADVERSE EVENTS:
Time Frame: AEs were recorded continuously starting from the signing of the ICF through the Study Termination visit, in those subjects who received at least one dose of Sci-B-Vac™, approximately 13 months.
Description: AEs were recorded continuously starting from the signing of the ICF through the Study Termination visit, in those subjects who have been actually dosed.
Arm/Group | Sci-B-Vac™
All-Cause Mortality (participants affected / at risk) | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 76/91
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sci-B-Vac™ (N=91)
Headache (Nervous system disorders) | 34 (65)
Oropharyngeal pain (Gastrointestinal disorders) | 28 (39)
Rhinitis (Infections and infestations) | 27 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (18)
Pyrexia (General disorders) | 15 (18)
Asthenia (General disorders) | 12 (13)
Diarrhea (Gastrointestinal disorders) | 10 (11)
Toothache (Gastrointestinal disorders) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT04179786/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT04179786/SAP_001.pdf